CLINICAL TRIAL: NCT00727519
Title: A Randomized Clinical Trial for Estimating the Effects of Pomegranate Juice Consumption by Hemodialysis Patients on Oxidative Stress, Infections, Cardiovascular Events and Mortality
Brief Title: The Effect of Pomegranate Juice on Oxidative Stress in Hemodialysis Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Prof. Batya Kristal, Western Galilee Hospital-Nahariya
Purpose: Prevention
Other Study IDs: PJHD-23-7-08CTIL
Record Dates: First submitted 2008-07-27; First posted 2008-08-04 (Estimated); Last update posted 2010-03-23 (Estimated); Status verified 2010-03

CONDITIONS: End Stage Renal Disease; Hemodialysis
Keywords: Hemodialysis; Nephrology; Pomegranate Juice; Israel
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PG (Experimental)
  Interventions: Dietary Supplement: Pomegranate juice
- PL (Experimental)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Pomegranate juice
  Arms: PG
Dietary Supplement: Placebo
  Arms: PL

SUMMARY:
Pomegranate juice (PJ) consumption by hemodialysis patients will reduce the oxidative stress and the incidence of infections, cardiovascular events and mortality.

DETAILED DESCRIPTION:
The mortality rate in patients with end stage renal failure is substantially higher than in the general population, and deaths are mainly attributable to cardiovascular diseases and infections. There is accumulating evidence that supports the role for oxidative stress in damaging the immune system and in the pathogenesis of cardiovascular diseases in hemodialysis patients, therefore antioxidative treatment, which will reduce oxidative stress, may be beneficial.

Pomegranate juice contains antioxidants such as soluble polyphenols, tannins and anthocyanins and was shown to have anti-inflammatory, anti- bacterial and anti-atherosclerotic properties in mice and humans. However,the effects of pomegranate juice on oxidative stress, infections and cardiovascular events in hemodialysis patients are still not documented.

This is a randomized preventive intervention trial on hemodialysis patients from one dialysis centre in Israel. The patients will be enrolled and randomized to receive pomegranate juice or placebo. Patients will be followed for one year. The objective of this study is to investigate the effects of pomegranate juice (PJ) consumption by hemodialysis patients on the changes in oxidative stress and the incidence of infections, cardiovascular events and mortality.

ELIGIBILITY:
Inclusion Criteria:

* End Stage Renal Disease, stable chronic hemodialysis > 3 months
* Informed Consent.
* Man and women over 18 years.

Exclusion Criteria:

* Hemodialysis < 3 months
* Participation in other clinical trial
* Not eligible according to physician decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2008-07; Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Western Galilee hospital, Nahariya, Israel, Israel

REFERENCES:
- [Derived] Shema-Didi L, Kristal B, Sela S, Geron R, Ore L. Does Pomegranate intake attenuate cardiovascular risk factors in hemodialysis patients? Nutr J. 2014 Mar 4;13:18. doi: 10.1186/1475-2891-13-18. PMID 24593225